CLINICAL TRIAL: NCT01124513
Title: A Prospective Study of Melanin Index in Those With Fitzpatrick Skin Phototypes I-VI
Brief Title: Melanin Index in Those With Fitzpatrick Skin Phototypes I-VI
Acronym: Melanin Index
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, June Robinson, Professor of Dermatology, Northwestern University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: JR-STU27549
Record Dates: First submitted 2010-05-10; First posted 2010-05-17 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Erythema
Keywords: Melanin Index; Fitzpatrick Skin Phototype; Videodermoscopy; Spectrophotometry
MeSH Terms: conditions — Erythema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Digital Camera (Active Comparator): Digital camera images will be taken of a a 2cm^2 area of sun protected skin.
  Interventions: Procedure: Induced Erythema
- Spectrophotometer (Active Comparator): The probe of the protable reflectance spectrophotometer is lightly applied to the sufance of the skin and a reading is taken.
  Interventions: Procedure: Induced Erythema
- Videodermoscopy (Active Comparator): The instrument is put in contact with sun protected skin and an image is taken of a 2 cm^2 area.
  Interventions: Procedure: Induced Erythema

INTERVENTIONS:
Procedure: Induced Erythema — Study personnel will induce erythema by sequentially applying ice for approximately 2 minutes to the 2 cm^2 target region of the upper volar arm. This erythema is a reaction to the vasoconstriction caused by skin cooling. The vasoconstriction is visually monitored to determine the onset of the vascular dilation that occurs after cessation of cooling. Images with the Digital Camera, Spectrophotometer and Videodermoscope are re-taken.

SUMMARY:
The "gold standard" method of assessing skin pigmentation is spectrophotometry; however, even as early as 1961 the potential for confounding by dilatation of blood vessels was recognized. (Monash 1961) Manual compression was used to express the blood from the field being measured. The red reflectance captured by reflectance spectrophotometer introduced an uncontrollable variable when measuring the tanning /pigmentation response of skin tone/color. Room temperature induced increased or decreased blood flow through the skin, which altered the findings by spectrophotometer. Other potentially confounding variables that changed blood flow were: recent exercise, and the flushing/blushing for emotional reasons. Since these conditions were difficult to reliably control on the sun exposed extremities, spectrophotometry was not a practical method to assess change in melanin over time as an outcome measure for efficacy of sun protection.

Digital imaging with videodermatoscopy utilizing a portable device that is supported by a laptop computer, provides a high resolution digital image for analysis. (EasyScan) As described by Yamamoto et al (2008), applying the Image J freeware to quantify the pigmentation in the digital image holds promise as a practical objective method to reliably assess skin tones based on the melanin content in a non invasive manner. With standardization, the software and hardware may quantify the constitutive pigment in the sun protected skin as the melanin index.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* fluent in English
* able to complete the study procedures including answering questionnairs
* willing to apply ice to left upper inner arm
* willing to have digital photos, dermatoscopic photos and spectrophometry readings taken of left upper inner arm

Exclusion Criteria:

* have a history of vitiligo or currently has vitiligo
* use self-tanning products or tan accelerators ont he left upper inner arm int he 4 weeks prior to enrollment
* history of cold urticaria or conenctive tissue disease such as scleroderma

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2010-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Change in Melanin Index | 2 minutes
  Compare the MI obtained by the digital camera, videodermoscope and spectrophotmetry between the usual conditions and after the induction of erythema.
Change in Melanin Index for 3 methods (digital camera, videodermoscope and spectrophotmetry) vs. patient-reported skin type vs. dermatologist-determined skin type | Up to 10 minutes
  Correlate the melanin index under usual conditions by each of the 3 methods (digital camera, videodermoscope and spectrophotometry) with the Fitzpatrick skin phyototype as determined by the patients' responses to standard questions, and the dermatologist's determination of skin type.
Difference in Time to Complete each of the 3 methods (digital camera, videodermoscope and spectrophotometer) | Up to 10 minutes
  Compare the time of testing (duration of each test for thes ubject, time spent by the research assistant administering the test) between the digitical camera, videodermoscope and spectrophotometer.
Desirability and Relevance of Videodermoscopy Image | Up to 10 minutes
  Assess desirability and relevance of the image obtained by videodermoscopy to the subject especially with reference to the subject's assessment of their risk of sunburning.

CONTACTS AND LOCATIONS:
Overall Officials: June K Robinson, MD, Principal Investigator — Northwestern University; Dennis P West, PhD, Study Director — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Result] Eilers S, Bach DQ, Gaber R, Blatt H, Guevara Y, Nitsche K, Kundu RV, Robinson JK. Accuracy of self-report in assessing Fitzpatrick skin phototypes I through VI. JAMA Dermatol. 2013 Nov;149(11):1289-94. doi: 10.1001/jamadermatol.2013.6101. PMID 24048361